CLINICAL TRIAL: NCT01817972
Title: A Phase III, Randomized, Double-blind Trial in the Comparison of Cimzia Versus Cimzia Plus Azathioprine in the Change in Mean SES-CD (Simple Endoscopic Scores-Crohn's Disease) Scores in the Treatment of Active, Moderate to Severe Crohn's Disease
Brief Title: Cimzia Versus Cimzia Plus Azathioprine in the Treatment of Active Crohn's Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gastroenterology Research of America (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CP-GAME01; Randall 2010-02 (Other Grant/Funding Number: UCB Inc.)
Record Dates: First submitted 2013-03-19; First posted 2013-03-26 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2013-03

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Crohn's colitis; Crohn's ileocolitis
MeSH Terms: conditions — Crohn Disease | interventions — Certolizumab Pegol; Azathioprine; Adenosine Triphosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Certolizumab pegol-Placebo Azathioprine (Placebo Comparator): Certolizumab pegol (Cimzia) 400mg Subcutaneous injection (per standard induction protocol) - which is at week 0, week 2, week4, week 6, then every 4 weeks until week 26. You will also be receiving Azathioprine placebo tablets at a dosage of 1.5mg per kilogram of body weight once a day for 26 weeks. They will be 50mg tablets. This is not active Azathioprine.
  Interventions: Biological: Certolizumab pegol
- Certolizumab pegol plus Azathioprine (Active Comparator): Certolizumab pegol (Cimzia) 400mg Subcutaneous injection (per standard induction protocol) - which is at week 0, week 2, week4, week 6, then every 4 weeks until week 26. You will also be receiving Azathioprine tablets at a dosage of 1.5mg per kilogram of body weight once a day for 26 weeks. They will be 50mg tablets.
  Interventions: Biological: Certolizumab pegol; Drug: Azathioprine

INTERVENTIONS:
Biological: Certolizumab pegol — Subcutaneous injection
  Other Names: Cimzia
Drug: Azathioprine — 50mg tablets
  Other Names: Imuran, Azasan, generic Azathioprine
  Arms: Certolizumab pegol plus Azathioprine

SUMMARY:
This is a randomized, double blind trial of combination therapy (Cimzia plus Azathioprine) versus mono therapy (Cimzia alone) and the improvement in mean SES-CD (Simple Endoscopic Scoring in Crohn's Disease) score.

It is a trial where the investigators are administering biological therapy by itself and biological therapy plus an immunosuppressive medicine in combination to see which form of therapy has a better effect on healing ulcerations in the small intestine and colon that are due to a flare up of Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has signed an Informed Consent Form (ICF).
2. The patient is ambulatory, community-dwelling male or non-pregnant female and is aged between 18 and 70 years at the Screening Visit. Lactating females must agree not to breastfeed.
3. Sexually active female patients of childbearing potential must agree to use one of the following methods of birth control from the date they sign the ICF until the conclusion of the trial:

   a. Hormonal contraception (i.e. oral contraceptive, contraceptive implant, or injectable hormonal contraceptive) b. Double-barrier birth control (e.g. condom plus intrauterine device, diaphragm plus spermicide) c. Surgical sterilization (i.e. bilateral oophorectomy, hysterectomy, or tubal ligation) d. Maintenance if a monogamous relationship with a male partner who has been surgically sterilized by vasectomy
4. Females of childbearing potential must have a negative serum pregnancy test at the Randomization Visit (first study treatment visit) prior to dosing.
5. Patient has no clinically significant findings on a physical examination, 12-lead electrocardiogram (ECG) and clinical laboratory tests (clinical chemistry panel, complete blood count [CBC], urinalysis [UA]) after signing the ICF but before receiving the first dose of study drug. (Note: The Investigator will determine if a particular finding is clinically significant. In making this determination, the investigator will consider whether the particular finding could prevent the patient from performing any of the protocol-specified assessments, could represent a condition that would exclude the patient from the trial, could represent a safety concern if the patient participates in the trial, or could confound the trial-specified assessments of safety or efficacy.)
6. Patient is fluent in English.
7. Are considered eligible according to the following TB screening criteria:

   • Have no history of latent or active TB prior to screening. An exception is made for patients with a history of latent TB and documentation of having completed appropriate treatment for latent TB within 3 years prior to the first administration of study agent. Appropriate documentation to verify that there had been treatment with a antituberculous treatment must be established prior to study participation.

   • Have no signs or symptoms suggestive of active TB upon medical history and/or physical examination.

   • Have no recent close contact with a person with active TB.

   • Subject has a negative purified protein derivative test within 30 days prior to the first dose. Tuberculin skin tests should be considered positive when they have greater than or equal to 5 mm of induration at 48 to 72 hours after test is placed. Subjects with a positive tuberculin skin test (if less than or equal to 14 mm of induration) are allowed if they have a history of Bacillus Calmette-Guerin vaccination with a negative Quantiferon test in the past year, no symptoms per tuberculosis workup, and a negative chest X-ray.
8. Be able to adhere to the required study visit schedule and comply with noted protocol requirements.
9. Subject has established ileal, ileo-colonic, or colonic Crohn's disease for a minimum of 3 months.
10. Subject has moderately to severely active Crohn's disease, as defined by a Crohn's Disease Activity Index (CDAI) score from 225 to 450 at screening and baseline and must also have an SES score that falls under the auspice of moderate to moderately severe disease (10-15).
11. Subject has evidence of active inflammation, as demonstrated by any of the following:

    * Elevated C reactive protein (CRP) at screening (>2.87 mg/L, or upper limit of normal (ULN) as set by local laboratory)
    * Endoscopic evidence of inflammation during the screening period or within 8 weeks prior to the screening period
12. Subjects are allowed to continue on concurrent treatment with the following agents:

    * 5-aminosalicylates, if stable dosage for at least 2 weeks prior to screening (same dosage to be maintained throughout the trial)
    * Probiotics, provided that the dose has been stable for the 2 weeks prior to enrollment
    * Antidiarrheals (eg, loperamide, Imodium) for control of chronic diarrhea; as per standard CDAI protocols, the use of antidiarrheals will be assessed at each visit.

Additional eligibility information

SES-CD The subject has a diagnosis of active moderate to severe CD at screening with these specific findings: the presence of large ulcerations (0.5cm is the minimal diameter in size to be categorized as large - this also constitutes between 2-3 points on the SES-CD score), the extent of ulcerated surface (the minimal percentage has got to be at least 10% - this also constitutes between 2-3 points on the SES-CD score), the extent of the affected surface (50% is the minimal percentage to fall in the moderate category - would constitute between 2-3 points on the SES-CD score) and finally the presence and type of narrowing found (number of strictures found and if the colonoscope can be passed or cannot be passed - this also constitutes between 2-3 points on the SES-CD score). The minimal score will be between 10 and 15. The local endoscopist (investigator) will determine whether subjects meet the entrance criteria from the SES scoring perspective. An appendix will be attached to define in a table the simple endoscopic scoring for Crohn's Disease (Appendix 1).

CDAI Crohn's Disease Activity Index scoring: this consists of eight variables including five subject reported outcomes. Variables 1,2,3,4 and 5 will be obtained from the patient's diary (see table 2a, subject diary, under Appendix 2, Crohn's Disease Activity Index Variables) completed by the patient during the 7 days prior to each CDAI evaluation. The Standard Height and Weight Table (Table 2b) must be used to calculate variable 8. The score from each variable is weighted by applying the multiplier shown. The total CDAI score is then determined by calculating the sum of the individual, weighted scores. A minimum score of 225 points is required and cannot exceed 450. These are the two primary criteria for entry that have to do with the study outcomes proposed.

Exclusion Criteria:

1. The patient has any condition, including clinically significant abnormalities on Screening laboratory test and/or medical history found during Screening assessments, or any acute or chronic condition, that, in the opinion of the investigator, constitutes a risk for the patient or a contraindication for participation in and completion of the study, or could interfere with study objectives, conduct, or evaluations (such as unstable diabetes mellitus, thyroid disease, vascular disease, end-stage coronary disease, pulmonary disease, liver disease, renal disease and any metabolic disorders that are also uncontrolled).
2. The patient has major surgery scheduled during the study period.
3. The patient has a history of cancer, except for adequately treated basal cell carcinoma of the skin, cervical dysplasia, or carcinoma in situ of the skin or the cervix.
4. Are pregnant, nursing, or planning pregnancy (both men and women) during the trial or for a 6-month period thereafter.
5. Have shown a previous immediate hypersensitivity response, including anaphylaxis, to an immunoglobulin product (plasma-derived or recombinant, e.g. monoclonal antibody).
6. Have received within 3 months prior to screening or are expected to receive any live viral (e.g. small-pox) or live bacterial vaccinations during the trial or up to 3 months after the last administration of study agent.
7. Have evidence of an active infection at the time of randomization or have had a serious infection not related to CD (e.g., hepatitis, pneumonia, or pyelonephritis), within 6 months prior to screening.
8. Have or have had an opportunistic infection (e.g., herpes zoster [shingles], cytomegalovirus, Pneumocystis carinii, aspergillosis, histoplasmosis, or mycobacteria other than TB) within 6 months prior to screening. Have current active hepatitis B (including chronic active hepatitis B or asymptomatic carrier state [hepatitis B surface antigen positive; HBsAg-positive]) or a history of hepatitis C infection.
9. Chronic pancreatitis.
10. Have any condition that, in the opinion of the investigator, would compromise the well-being of the patient or the study or prevent the patient from meeting or performing study requirements.
11. Have multiple sclerosis or other central demyelinating disorder.
12. Have a history of lymphoproliferative disease including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy of unusual size or location (e.g., nodes in the posterior triangle of the neck, intraclavicular, epitrochlear, or periaortic areas), or splenomegaly.
13. Have a transplanted organ (with the exception of a corneal transplant performed > 3 months prior to screening).
14. Have documented or suspected human immunodeficiency virus (HIV) infection.
15. Evidence of abdominal abscess at the initial screening visit
16. Extensive colonic resection, subtotal or total colectomy
17. History of >3 small bowel resections or diagnosis of short bowel syndrome
18. Have received tube feeding, defined formula diets, or parenteral alimentation within 21 days prior to the administration of the first dose of study drug
19. Ileostomy, colostomy, or known fixed symptomatic stenosis of the intestine
20. Within 30 days prior to enrollment, have received any of the following for the treatment of underlying disease:

    * Non-biologic therapies (e.g., cyclosporine, thalidomide)
    * A non-biologic investigational therapy
    * An approved non-biologic therapy in an investigational protocol

20. Within 60 days prior to enrollment, have received any of the following:

* Infliximab
* Certolizumab pegol
* Adalimumab
* Any other investigational or approved biological agent, other than local injections for non inflammatory bowel disease (IBD) conditions (e.g. intraocular-injections for the treatment of wet macular degeneration) 21. Any prior exposure to natalizumab, efalizumab, or rituximab 22. Evidence of or treatment for C. difficile infection or other intestinal pathogen within 28 days prior to enrollment 23. Have a history of substance abuse (drug or alcohol) within the previous 3 years, history of noncompliance to medical regimens, or other condition/circumstance that could interfere with the patient's adherence to protocol requirements (e.g., psychiatric disease, lack of motivation, travel, etc).

  24. Have Ulcerative Colitis as their diagnosis 25. Are employees of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-06 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Change in mean simple endoscopic scoring achieved by monotherapy versus combination therapy | At the beginning of the study and at week 27 of the study
  The primary objective is to compare the change in mean SES-CD score achieved by combination therapy (Cimzia plus AZP) versus mono therapy (Cimzia alone). A colonoscopy will be performed at the beginning of the trial and at the conclusion of the treatment period to see if there were any changes between the two treatment groups.

SECONDARY OUTCOMES:
Assess differences in response rates and remission rates between the two groups | At week 27 of the study which is their end of treatment study visit
  The secondary efficacy objective is to assess differences in response rates (which we will define for this trial as a drop to ≤10 on SES scoring)between the two groups.
Assess differences in response rates and remission rates between the two groups | At week 34 end of study
  The secondary efficacy objective is to assess differences in remission rates (no mucosal ulcerations at study end) between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Charles W Randall, MD, Principal Investigator — Gastroenterology Research of America; Carlo M Taboada, MD, Study Director — Gastroenterology Research of America
Locations (1):
- Gastroenterology Research of America, San Antonio, Texas, United States